CLINICAL TRIAL: NCT00315588
Title: Islet Cell Transplantation in Patients With Type I Diabetes With Previous Kidney Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rodolfo Alejandro (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Diabetes Research Institute Foundation (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Rodolfo Alejandro, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000/0329; 5R01DK055347 (NIH); 5R01DK025802 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Islet Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Islet Transplantation (Experimental): Islet Transplantation in subjects with a previous kidney transplant.
  Interventions: Drug: Islet Transplantation

INTERVENTIONS:
Drug: Islet Transplantation — Islet Transplantation in subjects with a previous kidney transplant.
  Other Names: islet

SUMMARY:
The purpose of this study is to reverse hyperglycemia and insulin dependency, by islet cell transplantation, in patients with type 1 diabetes mellitus who have a stable kidney allograft.

DETAILED DESCRIPTION:
1. To reverse hyperglycemia and insulin dependency by islet cell transplantation, in patients with Type 1 Diabetes Mellitus who have a stable kidney allograft;
2. To eliminate the incidence of hypoglycemic coma and unawareness by islet cell transplantation;
3. To assess long-term function of successful islet cell transplants;
4. To determine whether the natural history of the microvascular, macrovascular and neuropathic complications of Diabetes Mellitus are altered following successful transplantation of islet cells.
5. To assess the effect of exenatide to improve islet graft function and survival in subjects that demonstrate partial graft loss and have returned to using exogenous insulin.
6. To assess the ability of exenatide to improve islet survival at time of islet transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 60 years of age.
2. Patients with type 1 diabetes mellitus.
3. Patients with a renal transplant that is more than 6 months old.
4. Patients with stable renal graft function for the preceding 6 months, i.e. no episodes of rejection and changes in serum creatinine no more than 0.5 mg/dl from baseline.
5. Patients who are taking tacrolimus, sirolimus +/- steroids for maintenance immunosuppression for at least 6 months and are tolerating levels satisfactory for islet transplantation without severe complications.
6. Patients with a body mass index (BMI) of less than or equal to 26.

Exclusion Criteria:

1. Stimulated or basal C-peptide > 0.3 ng/ml.
2. Patients with unstable renal function - serum creatinine greater than 0.5 mg/dl above baseline.
3. Patients with proteinuria (albuminuria > 300 mg in 24 hours +/- protein) of new onset since kidney transplantation. If proteinuria or albuminuria is thought to originate from the native kidney(s) this will not be an exclusion criterion.
4. Patients with corrected creatinine clearance of less than 40.
5. Patients weighing more than 80 kg.
6. Patients with a body mass index (BMI) of greater than 26.
7. Insulin requirement > 1.0 U/kg/d.
8. Anemia (hemoglobin: males < 11.0 g/dl; females < 10.0 g/dl).
9. Abnormal liver function tests (consistently > 1.5 x normal range).
10. Unstable diabetic retinopathy.
11. Evidence of acute or chronic active Epstein-Barr virus (EBV) infection (IgM ≥ IgG). Patients will be eligible if serological testing becomes consistent with previous exposure (i.e. IgG > IgM).
12. Patients with history of malignancy or current malignancy other than non-melanomatous skin cancer, or finding of any lesions or symptoms during screening that are suspicious for malignancy, until properly investigated and ruled out.
13. Patients with elevation of prostate-specific antigen > 4 unless malignancy has been excluded.
14. Patients with unstable cardiovascular status.
15. Patients with active infections until adequately treated, unless treatment is not judged as necessary by the investigators (including, but not limited to, mild skin and nail fungal infections).
16. Patients with serological evidence of infection with HIV, human t cell lymphotropic virus 1 (HTLV 1), HTLV 2, or hepatitis B (patients with serology consistent with previous vaccination and a history of vaccination are acceptable).
17. Patients with history and/or serological evidence of hepatitis C (those patients with hepatitis C, already transplanted in this protocol will continue in this trial).
18. Positive tuberculin test (unless proof of adequate treatment for latent tuberculosis can be provided).
19. Patients with active peptic ulcer disease, gallstones, hepatic hemangioma, or portal hypertension.
20. Patients who are pregnant or breastfeeding, or who intend to procreate.
21. Patients who are sexually active females who are not:

    * post-menopausal,
    * surgically sterile, or
    * using an acceptable method of contraception (oral contraceptives, Norplant, Depo-Provera, and barrier devices combined with spermicidal gel are acceptable; condoms used alone are not acceptable).
22. Active alcohol or substance abuse; smoking in the last 6 months.
23. Patients with evidence of sensitization, i.e. panel reactive antibody (PRA) testing greater than 20%.
24. Lack of updated immunizations per current Centers for Disease Control (CDC) guidelines, as well as immunization against hepatitis B, pneumococcus, and influenza (during season), unless medically contraindicated.
25. Patients with psychogenic factors, which are judged at psychological evaluation, which make it unsafe to undergo islet transplantation, or which preclude therapeutic compliance.
26. Patients with any condition or any circumstance that would make it unsafe to undergo an islet transplant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2000-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodolfo Alejandro, M.D., Principal Investigator — University of Miami
Locations (1):
- Diabetes Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cure P, Pileggi A, Froud T, Messinger S, Faradji RN, Baidal DA, Cardani R, Curry A, Poggioli R, Pugliese A, Betancourt A, Esquenazi V, Ciancio G, Selvaggi G, Burke GW 3rd, Ricordi C, Alejandro R. Improved metabolic control and quality of life in seven patients with type 1 diabetes following islet after kidney transplantation. Transplantation. 2008 Mar 27;85(6):801-12. doi: 10.1097/TP.0b013e318166a27b. PMID 18360260
- [Derived] Faradji RN, Froud T, Messinger S, Monroy K, Pileggi A, Mineo D, Tharavanij T, Mendez AJ, Ricordi C, Alejandro R. Long-term metabolic and hormonal effects of exenatide on islet transplant recipients with allograft dysfunction. Cell Transplant. 2009;18(10):1247-59. doi: 10.3727/096368909X474456. PMID 20003758
- [Derived] Tharavanij T, Betancourt A, Messinger S, Cure P, Leitao CB, Baidal DA, Froud T, Ricordi C, Alejandro R. Improved long-term health-related quality of life after islet transplantation. Transplantation. 2008 Nov 15;86(9):1161-7. doi: 10.1097/TP.0b013e31818a7f45. PMID 19005394
- See also: Research into finding the cure for types 1 and type 2 diabetes. — http://www.diabetesresearch.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Islet Transplantation: Islet transplantation in subjects with previous kidney transplant.
Period: Overall Study
Arm/Group | Islet Transplantation
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Insulin Independence.
Description: Number of Participants who Achieved Insulin Independence at 1 Year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 7
Participants | 2

2. Secondary Outcome: Stimulated C-peptide Greater Than 0.5 ng/ml
Description: Partial graft function, as evidenced by basal C-peptide greater than 0.5 ng/ml
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 7
Participants | 6

3. Secondary Outcome: Reduction of Insulin Requirements
Description: Reduction in insulin requirements in those patients who do not achieve insulin independence
Time Frame: 1year
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 5
Participants | 4

4. Secondary Outcome: Reduction in Severe Hypoglycemia, Improvement in Hypoglycemia Awareness
Description: Elimination or reduction in the incidence of hypoglycemic coma or unawareness
Time Frame: 1 years
Measure: Count of Participants; unit: Participants
Arm/Group | Islet Transplantation
Number analyzed (Participants) | 7
Participants | 6

ADVERSE EVENTS:
Arm/Group | Islet Transplantation
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplantation (N=7)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Chest Pain (Cardiac disorders) | 1 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Increased Serum Creatinine (Renal and urinary disorders) | 1 (1)
Limb edema (Vascular disorders) | 1 (1)
Squamous Cell Carcinoma in situ (Skin and subcutaneous tissue disorders) | 2 (2)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3)
Pneumonia (Infections and infestations) | 2 (2)
Head Injury (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Transplantation (N=7)
Tremors (Nervous system disorders) | 1 (5)
Insomnia (Nervous system disorders) | 2 (5)
Depression (Nervous system disorders) | 1 (2)
Memory loss (Nervous system disorders) | 1 (1)
Headaches (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (5)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Buccal ulcers (Gastrointestinal disorders) | 3 (5)
Acne/Folliculitis (Skin and subcutaneous tissue disorders) | 1 (3)
Rash (legs) (Skin and subcutaneous tissue disorders) | 1 (1)
Necrobiosis lipodica (Skin and subcutaneous tissue disorders) | 1 (1)
Onychomyosis (Skin and subcutaneous tissue disorders) | 1 (1)
Squamous cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (2)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
1st and 2nd degree burn (Skin and subcutaneous tissue disorders) | 1 (1)
Skin desquamation right index finger (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia Areata (Skin and subcutaneous tissue disorders) | 1 (1)
Onychocriptosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin, cracks on fingers (Skin and subcutaneous tissue disorders) | 1 (1)
Facial Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Increase creatinine (Renal and urinary disorders) | 2 (2)
Microalbuminuria (Renal and urinary disorders) | 3 (3)
Overt albuminuria (Renal and urinary disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Nausea and Vomiting (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
Bezoar (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Cholelithiasis (Gastrointestinal disorders) | 1 (1)
Intrahepatic Biliary dilation (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3)
Otitis Media (Infections and infestations) | 1 (1)
Dental Infection (Infections and infestations) | 1 (1)
Urinary Tract infection (Infections and infestations) | 3 (4)
EBV (Infections and infestations) | 2 (3)
Lower leg infection (Infections and infestations) | 1 (1)
Arthralgia/arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Low Extremity Edema (Blood and lymphatic system disorders) | 2 (2)
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Upper Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nodular Opacity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye surgery (Eye disorders) | 1 (1)
Blurred Vision (Eye disorders) | 2 (2)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Increased LFT (Gastrointestinal disorders) | 3 (3)
Ovarian Cyst (Reproductive system and breast disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes